CLINICAL TRIAL: NCT07356583
Title: Neonatal Enterovirus Infections in Italy: Virological Characterization, Genomic and Clinical-epidemiological Insights on Echovirus 11
Acronym: Entero-Neo
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other); Università di Genova, Genova (Unknown)
Responsible Party: Principal Investigator, Antonio Piralla, PhD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Entero-neo
Record Dates: First submitted 2025-12-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Enterovirus; Clinical Syndrome; Respiratory Complications; Gastrointestinal; Sepsis
Keywords: Enterovirus, E-11, NGS
MeSH Terms: conditions — Enterovirus Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Enterovirus genus, belonging to the Picornaviridae family, consists of positively polarized single-stranded RNA viruses classified into the species Enterovirus (EV, comprising Coxsackievirus, Echovirus and Poliovirus) A-J and Rhinovirus (RV) A-C, of which more than 200 different genotypes have been described. Enteroviruses have a global spread and are a common cause of febrile, gastroenteric and exanthematous diseases, usually self-limiting, which are widespread in infants and pediatric populations. However, they can occasionally cause serious diseases, including meningoencephalitis, myelitis, paralysis, myocarditis, sepsis, severe respiratory syndromes, and acute hepatitis. They can be transmitted by respiratory route, with most cases in temperate regions occurring during summer and early autumn. Enteroviruses are characterized by a rapid evolution determined by the high mutation rate (due to the presence of an RNA-dependent RNA-polymerase that lacks proofreading activity) and the high probability of undergoing recombination events. The latter, in particular inter-typical recombination, plays a crucial role in the evolutionary process of Enteroviruses and has been recognized as a major cause of the emergence of strains with higher pathogenicity and/or epidemic potential, although the associated genetic determinants are not known to date. Between July 2022 and April 2023, nine cases of neonatal Echovirus 11 (E-11) infection with severe liver failure and neurological and myocardial involvement were reported in France; seven of these cases resulted in fatal outcomes. Following these reports, the World Health Organization (WHO) issued an alert that quickly led to the identification of further cases in Italy, Spain, Croatia and the United Kingdom. As EV infections are not subject to systematic surveillance, there is a lack of data on the actual burden of disease associated with these infections. Thus, EV infections are underestimated and, even more so, data on their typing are scarce - if not absent -, which involve second-level analyses that are generally not carried out routinely in clinical microbiological diagnostic laboratories, are rarely available and are not systematically collected, not even at European level. A condition that therefore makes it impossible to estimate either the impact of EV infections in general, and of E-11 in particular, or the risk factors related to the most serious cases and the most significant transmission routes. Moreover, the characteristics of the immunological and inflammatory response to infection remain to be defined. These elements would allow, if available, the formulation of a specific case definition to ensure rapid laboratory confirmation and recognition of the disease.To strengthen knowledge of the spread and impact of enterovirus infections in newborns, with a focus on E-11, by carrying out the following activities, within the scope of the project's proposed objectives: design and pilot implementation (proof of concept) of epidemiological and genomic surveillance systems with potential national application; molecular characterization and evaluation of viral pathogenic features; search for possible immunological markers and host risk factors associated with severe EV disease, including E-11.

Specific objectives

1. To implement and validate a protocol for screening activities in neonatal units and neonatal intensive care units aimed at checking for the presence of infections caused by EV and identifying severe forms of infection, with particular attention to E-11.
2. Characterize EV strains, identified within the activities carried out by specific objectives 1, using next-generation sequencing (NGS) approaches to obtain the whole genome sequence and identify possible recombinant forms. Carry out phylogenetic analysis of the obtained sequences compared with those deposited in the main international databases, to define genomes that can be traced back to variant strains or with specific mutations in the genome.

ELIGIBILITY:
Inclusion Criteria:

Samples from consecutive neonates admitted to neonatal intensive care unit.

Exclusion Criteria:

Insufficient residual samples (volume less than 1 mL of nasal swab) will be excluded from the study

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates admitted to the neonatal intensive care unit.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of enteroviruses prevalence in neonates | From February 2026 to February 2027
  To strengthen knowledge of the spread and impact of enterovirus infections in newborns, with a focus on E-11, by carrying out the following activities, within the scope of the project's proposed objectives: design and pilot implementation (proof of concept) of epidemiological and genomic surveillance systems with potential national application; molecular characterization and evaluation of viral pathogenic features; search for possible immunological markers and host risk factors associated with severe EV disease, including E-11.
Neonatal enterovirus infections in Italy: virological characterization, genomic and clinical-epidemiological insights on Echovirus 11 | February 2026-February2027

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No